CLINICAL TRIAL: NCT04697277
Title: The Effect of Antibiotic Prophylaxis Timing on Intraoperative Nausea and Vomiting in Patients Undergoing Cesarean Section Under Regional Anesthesia.
Brief Title: Antibiotic Prophylaxis and Nausea and Vomiting in Cesarean Section Under Regional Anesthesia.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Bahattin Tuncali, Associate professor, MD, Baskent University Ankara Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KA15/197
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Intraoperative Nausea-retching-vomiting Episodes; Nausea Scores Will be Evaluated on the Verbal Analog Scale (VAS)
Keywords: antibiotic prophylaxis; nausea; vomiting; cesarean section; egional anesthesia
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A computer-generated random numbers table and sealed envelopes will be used to ensure randomization. The gynecologist performing the surgery, the anesthesiologist and the patients will not know the Group allocation. The medications will be prepared by the anesthesia technician responsible for the study. Prophylactic antibiotic and placebo will be prepared in 10 ml in the syringe and labeled as study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 (Prophylactic antibiotic 30 minutes before skin incision): Antibiotic diluted in 10 ml syringe 30 minutes before skin incision and after cord clamping, 0.9% NaCl in 10 ml syringe will be administered intravenously within 15 seconds.
  Interventions: Drug: Antibiotic prophylaxis timing (before skin incision and after cord clamping) for caesarean section
- Group 2 (Active Comparator): Group 2 (prophylactic antibiotic after cord clamping): 30 minutes before the skin incision, 0.9% NaCl in a 10 ml injector and after the cord is clamped, the antibiotic diluted in a 10 ml syringe will be administered intravenously within 15 seconds.
  Interventions: Drug: Antibiotic prophylaxis timing (before skin incision and after cord clamping) for caesarean section

INTERVENTIONS:
Drug: Antibiotic prophylaxis timing (before skin incision and after cord clamping) for caesarean section

SUMMARY:
The incidence of intraoperative nausea and vomiting in patients who undergo caesarean section (C/S) under regional anesthesia is approximately 30-80%. Hypotension, pain, visceral manipulation, fundal pressure, removal of the uterus during repair, intra-abdominal irrigation, central neural opioids, intravenous oxytocin and antibiotics are possible risk factors. Oxytocin and prophylactic antibiotics are administered simultaneously during C/S operation, especially after the umbilical cord is clamped. Simultaneous administration of drugs such as oxytocin and prophylactic antibiotics may induce nausea and vomiting after umbilical cord clamping in the patient. In this study, it was aimed to investigate the effect of prophylactic antibiotic administration 30 minutes before the incision and after cord clamping on intraoperative nausea and vomiting in patients undergoing elective C/S under regional anesthesia.

This study was planned to be carried out in Başkent University Zübeyde Hanım Research Center Operating Room with 120 pregnant women (≥ 37 gestational weeks) undergoing elective C/S under regional anesthesia in a prospective, randomized, double-blind manner.

Group 1 (Prophylactic antibiotic 30 minutes before skin incision): Antibiotic diluted in 10 ml syringe 30 minutes before skin incision and after cord clamping, 0.9% NaCl in 10 ml syringe will be administered intravenously within 15 seconds.

Group 2 (prophylactic antibiotic after cord clamping): 30 minutes before the skin incision, 0.9% NaCl in a 10 ml injector and after the cord is clamped, the antibiotic diluted in a 10 ml syringe will be administered intravenously within 15 seconds.

Intraoperative nausea-retching-vomiting episodes (0 = No symptoms, 1: Nausea (uncomfortable feeling with vomiting), 2: Gag (vomiting effort in which gastric contents cannot be expelled), 3: Vomiting (Gastric contents are forced by mouth. ejection)] will be recorded. Nausea scores will be evaluated on the verbal analog scale (VAS) with 11 points (0 = no nausea, 10 = the most severe nausea). Before anesthesia, all patients will be informed about the verbal analog scale (VAS) for nausea. VAS 1-3 = Mild Nausea, VAS 4-6 = Moderate nausea, VAS 7-10 = Severe nausea. Evaluations will be made at certain time intervals.

Before CSEA application Time interval between CSEA application and fetus discharge Time interval between fetus exit and expulsion of the uterus Time interval between expulsion of the uterus and insertion into the abdomen Time interval between insertion of the uterus in the abdomen and closing the fascia Time interval between fascia closure and skin closure Time interval between skin closure and patient transport to the recovery unit Nausea-retching-vomiting episodes, current systolic/diastolic blood pressure values, nausea-vomiting scores, antiemetic and / or ephedrine requirement, amount of intravenous fluid infused will be recorded.

Intraoperative prophylactic antibiotic use is considered as one of the possible causes of intraoperative nausea and vomiting in patients who underwent cesarean section under regional anesthesia. We believe that the results of our study can make contribution on both intraoperative nausea-vomiting etiology in cases undergoing cesarean section under regional anesthesia and the steps that can be taken to prevent it.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (≥ 37 gestational weeks) undergoing elective C/S under regional anesthesia

Exclusion Criteria:

* Emergency C/S cases
* Patients who had nausea before C/S
* Patients who used antiemetics within 24 hours before C/S
* Patients who have a history of smoking, postoperative nausea-vomiting, motion sickness, and hyperemesis before C/S
* Patients with history of diabetes, morbid obesity (Body Mass Index> 40) and gastrointestinal disease
* Psychiatric disorders
* Patients who are allergic to the drugs to be used in the study
* Patients for whom regional anesthesia is contraindicated

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women undergoing C/S under regional anesthesia
Enrollment: 120 (Estimated)
Dates: Start 2015-08-20 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative nausea-retching-vomiting episodes | Intraoperative
  0 = No symptoms, 1: Nausea (uncomfortable feeling with vomiting), 2: Gag (vomiting effort in which gastric contents cannot be expelled), 3: Vomiting (Gastric contents are forced by mouth. ejection)

SECONDARY OUTCOMES:
Nausea score | Intraoperative
  Nausea score will be evaluated on the verbal analog scale (VAS) with 11 points (0 = no nausea, 10 = the most severe nausea). Before anesthesia, all patients will be informed about the verbal analog scale (VAS) for nausea. VAS 1-3 = Mild Nausea, VAS 4-6 = Moderate nausea, VAS 7-10 = Severe nausea.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Balki M, Carvalho JC. Intraoperative nausea and vomiting during cesarean section under regional anesthesia. Int J Obstet Anesth. 2005 Jul;14(3):230-41. doi: 10.1016/j.ijoa.2004.12.004. PMID 15935649
- [Background] Fujii Y. Retraction Notice: Prevention of emetic episodes during cesarean delivery performed under regional anesthesia in parturients. Curr Drug Saf. 2007 Jan;2(1):25-32. doi: 10.2174/157488607779315381. PMID 18690947
- [Background] Hopkins L, Smaill F. Antibiotic prophylaxis regimens and drugs for cesarean section. Cochrane Database Syst Rev. 2000;(2):CD001136. doi: 10.1002/14651858.CD001136. PMID 10796247
- [Background] Costantine MM, Rahman M, Ghulmiyah L, Byers BD, Longo M, Wen T, Hankins GD, Saade GR. Timing of perioperative antibiotics for cesarean delivery: a metaanalysis. Am J Obstet Gynecol. 2008 Sep;199(3):301.e1-6. doi: 10.1016/j.ajog.2008.06.077. PMID 18771991
- [Background] Sullivan SA, Smith T, Chang E, Hulsey T, Vandorsten JP, Soper D. Administration of cefazolin prior to skin incision is superior to cefazolin at cord clamping in preventing postcesarean infectious morbidity: a randomized, controlled trial. Am J Obstet Gynecol. 2007 May;196(5):455.e1-5. doi: 10.1016/j.ajog.2007.03.022. PMID 17466699
- [Background] Thigpen BD, Hood WA, Chauhan S, Bufkin L, Bofill J, Magann E, Morrison JC. Timing of prophylactic antibiotic administration in the uninfected laboring gravida: a randomized clinical trial. Am J Obstet Gynecol. 2005 Jun;192(6):1864-8; discussion 1868-71. doi: 10.1016/j.ajog.2004.12.063. PMID 15970833
- [Background] Committee opinion no. 465: antimicrobial prophylaxis for cesarean delivery: timing of administration. Obstet Gynecol. 2010 Sep;116(3):791-792. doi: 10.1097/AOG.0b013e3181f68086. PMID 20733474
- [Background] Raghunathan K, Connelly NR, Friderici J, Naglieri-Prescod D, Joyce R, Prasanna P, Ponnusamy N. Unwarranted variability in antibiotic prophylaxis for cesarean section delivery: a national survey of anesthesiologists. Anesth Analg. 2013 Mar;116(3):644-8. doi: 10.1213/ANE.0b013e318276cf72. Epub 2013 Feb 11. PMID 23400990
- [Background] Jenkins JG, Khan MM. Anaesthesia for Caesarean section: a survey in a UK region from 1992 to 2002. Anaesthesia. 2003 Nov;58(11):1114-8. doi: 10.1046/j.1365-2044.2003.03446.x. PMID 14616600
- [Background] Voigt M, Frohlich CW, Huttel C, Kranke P, Mennen J, Boessneck O, Lenz C, Erbes T, Ernst J, Kerger H. Prophylaxis of intra- and postoperative nausea and vomiting in patients during cesarean section in spinal anesthesia. Med Sci Monit. 2013 Nov 14;19:993-1000. doi: 10.12659/MSM.889597. PMID 24226381
- [Background] Dasgupta M, Biswas BN, Chatterjee S, Mazumder P, Bhanja Chowdhury M. Randomized, placebo-controlled trial of granisetron for control of nausea and vomiting during cesarean delivery under spinal anesthesia. J Obstet Gynaecol India. 2012 Aug;62(4):419-23. doi: 10.1007/s13224-012-0291-0. Epub 2012 Oct 16. PMID 23904702
- [Background] Watcha MF. The cost-effective management of postoperative nausea and vomiting. Anesthesiology. 2000 Apr;92(4):931-3. doi: 10.1097/00000542-200004000-00007. No abstract available. PMID 10754609
- [Background] Koch KL, Frissora CL. Nausea and vomiting during pregnancy. Gastroenterol Clin North Am. 2003 Mar;32(1):201-34, vi. doi: 10.1016/s0889-8553(02)00070-5. PMID 12635417
- [Background] Manullang TR, Viscomi CM, Pace NL. Intrathecal fentanyl is superior to intravenous ondansetron for the prevention of perioperative nausea during cesarean delivery with spinal anesthesia. Anesth Analg. 2000 May;90(5):1162-6. doi: 10.1097/00000539-200005000-00030. PMID 10781472
- [Background] Demirhan A, Tekelioglu YU, Akkaya A, Ozlu T, Yildiz I, Bayir H, Kocoglu H, Duran B. Antiemetic effects of dexamethasone and ondansetron combination during cesarean sections under spinal anaesthesia. Afr Health Sci. 2013 Jun;13(2):475-82. doi: 10.4314/ahs.v13i2.39. PMID 24235952
- [Background] Griffiths JD, Gyte GM, Paranjothy S, Brown HC, Broughton HK, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007579. doi: 10.1002/14651858.CD007579.pub2. PMID 22972112
- [Background] Baaqeel H, Baaqeel R. Timing of administration of prophylactic antibiotics for caesarean section: a systematic review and meta-analysis. BJOG. 2013 May;120(6):661-9. doi: 10.1111/1471-0528.12036. Epub 2012 Nov 6. PMID 23126271
- [Background] Heesen M, Klohr S, Rossaint R, Allegaert K, Allegeaert K, Deprest J, Van de Velde M, Straube S. Concerning the timing of antibiotic administration in women undergoing caesarean section: a systematic review and meta-analysis. BMJ Open. 2013 Apr 18;3(4):e002028. doi: 10.1136/bmjopen-2012-002028. Print 2013. PMID 23604346
- [Background] Camann W, Tuomala R. Antibiotic prophylaxis for cesarean delivery: always before skin incision! Int J Obstet Anesth. 2011 Jan;20(1):1-2. doi: 10.1016/j.ijoa.2010.09.015. Epub 2010 Dec 3. No abstract available. PMID 21126866